CLINICAL TRIAL: NCT04961515
Title: A Phase II Study of Orelabrutinib, Sintilimab and Temozolomide in Treating Patients With Relapsed or Refractory Central Nervous System Lymphoma
Brief Title: Orelabrutinib, Sintilimab and Temozolomide in Relapsed or Refractory Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Wenzhou Central Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang Provincial Tongde Hospital (Other); First People's Hospital of Hangzhou (Other); Zhejiang Provincial People's Hospital (Other); Jinhua Central Hospital (Other); Jinhua People's Hospital (Other); Yinzhou Hospital Affiliated to Medical School of Ningbo University (Other); Huzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I2021001524
Record Dates: First submitted 2021-06-15; First posted 2021-07-14 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Primary Central Nervous System Hodgkin Lymphoma
MeSH Terms: interventions — orelabrutinib; sintilimab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OST regimen (Experimental): Participants will receive:
  1. Orelabrutinib: 150 mg orally once daily;
  2. Sintilimab: 200 mg intravenously every 3 weeks;
  3. Temozolomide: 150 mg/m² orally on days 1-5 of each 21-day cycle; Treatment consists of up to six 21-day cycles (induction phase), followed by sintilimab monotherapy maintenance until disease progression (PD), intolerable toxicity, investigator/patient decision to withdraw, or completion of 2 years total treatment (whichever occurs first). Tumor response will be assessed by MRI every two cycles during induction and quarterly thereafter
  Interventions: Drug: Orelabrutinib; Drug: Sintilimab; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib: 150 mg orally once daily
Drug: Sintilimab — Sintilimab: 200 mg intravenously every 3 weeks
Drug: Temozolomide (TMZ) — Temozolomide: 150 mg/m² orally on days 1-5 of each 21-day cycle

SUMMARY:
This phase II trial is evaluating the efficacy and side effect of orelabrutinib, sintilimab and temozolomide as possible treatments for relapsed or refractory central nervous system lymphoma.

DETAILED DESCRIPTION:
Orelabrutinib and anti-PD-1 monoclonal antibodies represent promising therapeutic classes for central nervous system lymphoma (CNSL). Given the poor outcomes and limited treatment options for relapsed or refractory CNSL, this study aims to evaluate the efficacy and toxicity of orelabrutinib combined with temozolomide and sintilimab in this population.

Participants will receive fixed-dose orelabrutinib, sintilimab, and temozolomide for up to six 21-day cycles (induction phase), followed by sintilimab maintenance until disease progression (PD), intolerable toxicity, investigator/patient decision to withdraw, or a maximum treatment duration of 2 years (whichever occurs first). Tumor response will be assessed by MRI every two cycles during induction and every three months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented primary central nervous system(CNS) lymphoma or secondary diffuse large B-cell lymphoma (DLBCL) isolated to CNS.
2. Relapsed or refractory disease with at least 1 prior methotrexate-based therapy
3. Participant must be able to understand and willing to sign a written informed consent document.
4. Participant must have signed and dated written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.
5. Participant must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study.
6. Participant must be at least 18 years old on day of signing informed consent.
7. PCNSL subjects should have evidence of measurable or evaluable enhancing disease on MRI
8. Able to submit at least 10 but up to 20 unstained formalin-fixed, paraffin-embedded (FFPE) slides from the initial or most recent tissue diagnosis for correlative studies. Histologically confirmed tissue will be required from the time of relapse or at the time of initial surgery. If tissue is unavailable and/or diagnosis was made from cerebrospinal fluid or vitreal biopsy, approval from the overall principal investigator is needed.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3.
10. Life expectancy of >3 months (in the opinion of the investigator)
11. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1
12. Must be able to tolerate lumbar puncture and MRI/CT.
13. Demonstrate adequate organ function as defined below, all screening labs should be performed within 14 days of treatment initiation.

    1. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
    2. Platelets ≥ 75 x 10^9/L and no platelet transfusion within the past 7 days prior to initiation of protocol treatment
    3. Prothrombin time (PT), partial thromboplastin time (PTT), and international normalized ratio (INR) < 2 times the upper limit of normal
    4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal
    5. Serum bilirubin ≤ 1.5 times the upper limit of normal
    6. Creatinine clearance > 30 mL/min calculated by the Cockcroft-Gault formula using actual body weight
14. Women of child-bearing potential, must agree to use a highly effective method of contraception consistently and correctly as described below during study treatment and for 120 days after study discontinuation.
15. Male participants must agree to use at least one of the following methods of contraception starting with the first dose of study therapy through 120 days after the last dose of therapy:
16. Ability to swallow oral medications.

Exclusion Criteria:

1. CNSL with systematic disease.
2. The pathological diagnosis was T-cell lymphoma.
3. Prior chemotherapy within 4 weeks or prior targeted small molecule therapy within 2 weeks , prior antibody-drug-conjugates within 10weeks, autologous stem cell transplant within 6 months, prior to the first day of study treatment, prior to the first day of study treatment.
4. Prior allogenic stem cell transplant.
5. Participation in another clinical study with an investigational product during the 4 weeks prior to the first day of study treatment.
6. External beam radiation therapy to the CNS within 14 days of the first day of study treatment.
7. Patient requires more than 8 mg of dexamethasone daily or the equivalent for control of CNS symptoms at the time of initiation of study therapy. Patients must taper off high dose corticosteroids for the control of CNS symptoms within 14 days after starting on study therapy.
8. History of intracranial hemorrhage or clinically significant stroke within 6 months prior to first day of study treatment
9. History of significant gastrointestinal disease that would limit absorption of oral medications.
10. Active concurrent malignancy requiring active therapy.
11. Prior therapy with a checkpoint inhibitor or BTK inhibitor.
12. Warfarin or any other Coumadin-derivative anticoagulant or vitamin K antagonists. Patients must be off warfarin-derivative anticoagulants for at least seven days prior to starting the study drug. Use of low molecular weight heparin and novel oral anticoagulants (eg. rivaroxaban, apixaban) is permitted if required.
13. Concurrent use of a moderate or strong inhibitor or inducer of the P450 isoenzyme CYP3A. Participants must be off P450/CYP3A inhibitors and inducers prior to starting the study drug.
14. Receipt of live attenuated vaccine within 30 days prior to the first day of study treatment. Note: Patients, if enrolled, should not receive live vaccine while receiving IP and up to 30 days after the last day of study treatment.
15. Suspicion of or confirmed progressive multifocal leukoencephalopathy
16. Active autoimmune disease (including autoimmune hemolytic anemia and immune thrombocytopenia purpura) requiring systemic treatment within the past two years (i.e. with the use of disease modifying agents, corticosteroids, or immunosuppressive drugs). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., due to Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
    6. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroids replacement therapy for adrenal or pituitary insufficiency, etc.)
17. Significant medical diseases or conditions, as assessed by the investigator, that would substantially increase the risk to benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction in the past 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, severely immunocompromised state, and congestive heart failure, New York Heart Association Class III-IV.
18. Known bleeding diathesis (e.g. von Willebrand's disease), hemophilia, or active bleeding.
19. Known Human immunodeficiency virus (HIV) infection.
20. Known active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests and/or PCR.
21. History of invasive fungal infection, including invasive aspergillosis, or known active tuberculosis.
22. Major surgery ≤ 6 weeks prior to starting the trial treatment (or has not recovered from the side effects of such surgery) or plans to have surgery within 2 weeks of the first dose of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2years
  The objective response rate (ORR) is defined as the proportion of patients with a best response of CR or PR

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival (OS) | 2 years
  OS is defined as the duration of time from start of treatment to time of death.
Duration of response | 2 years
  The duration of overall response is measured from the time measurement

OTHER OUTCOMES:
ctDNA mutation and mean ctDNA concentration in serum and cerebrospinal fluid | Baseline, every two months for up to three years after treatment
  Types of ctDNA mutations and frequency are measured by next generation sequencing. The mean ctDNA concentration is the concentration of ctDNA expressed as mean tumor molecules /ml at specific time points.
The levels of cytokine concentration in serum and cerebrospinal fluid | Baseline, every two months for up to three years after treatment
  The levels of cytokine will be analyzed by ELISA in all patients recruited. The cytokine profile includes IL-6, IL-10, TNF-α, IFN-γ, IL-2 and IL-4

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No